CLINICAL TRIAL: NCT02648256
Title: Pneumocystis Pneumonia Diagnosis in HIV- Patients: Assessment of the Real Time Polymerase Chain Reaction Quantification on Oropharyngeal Rinse
Brief Title: Pneumocystis Pneumonia Diagnosis in HIV- Patients
Acronym: PNEUMOQUANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-A00408-41; 35RC14_9890 (Other: Other Identifier)
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Pneumonia, Pneumocystis
Keywords: Pneumocystis jirovecii; Polymerase Chain Reaction; Oropharyngeal Rinse
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oropharyngeal rinse (Experimental): Polymerase Chain Reaction on Oropharyngeal rinse:
  Dosage of Pneumocystis jiroveci will be performed on the broncho-alveolar lavage following the usual routine diagnosis.
  Polymerase Chain Reaction will be performed on the broncho-alveolar lavage and the oropharyngeal rinse (not communicated to the clinician result) in the same series, in order to compare the results of the fungal quantification.
  Interventions: Other: Polymerase Chain Reaction on Oropharyngeal rinse

INTERVENTIONS:
Other: Polymerase Chain Reaction on Oropharyngeal rinse

SUMMARY:
Pneumocystis jirovecii pneumonia is a serious and frequent infection in immunocompromised patients, whose evolution is potentially fatal if untreated. It is the most common opportunistic infections classifying patients infected with human immunodeficiency virus (human immunodeficiency virus +) at the stage acquired immune deficiency syndrome. Data from the french Institute for Health Watch showed in 2011 that 31% of 1400 cases of acquired immune deficiency syndrome were revealed by Pneumocystis jirovecii pneumonia.

Pneumocystis jirovecii pneumonia also increasingly concerns immunocompromised human immunodeficiency virus negative patients, due to the increasing use of immunosuppressive therapies (including corticosteroids), of anticancer cytostatics and biotherapies, in the context of grafts, transplants, but also from autoimmune or inflammatory chronic diseases.

Recent data show that the number of cases occurring in patients Pneumocystis jirovecii pneumonia human immunodeficiency virus - in France is now higher than the cases occurring in Pneumocystis jirovecii pneumonia +. The severity of the Pneumocystis jirovecii pneumonia is increased in patients with human immunodeficiency virus -, in whom the evolution is faster, with mechanical ventilation often required and higher mortality, requiring a fast and early diagnosis. Routine diagnosis relies on the detection of the fungus in the bronchoalveolar lavage, using stains (May Grunwald Giemsa or immunofluorescence) and Polymerase Chain Reaction. Polymerase Chain Reaction provides a diagnostic gain in immunocompromised patients not infected with human immunodeficiency virus that may present a pejorative table quickly despite low fungal burden. However, the deoxyribonucleic acid of the fungus can sometimes be detected in the absence of scalable Pneumocystis jirovecii pneumonia, and then shows a pulmonary colonization by Pneumocystis jirovecii. It is therefore important to improve the positive predictive value of Pneumocystis Polymerase Chain Reaction, to guide the management of optimal patient.

In this work, the investigators propose to evaluate the Polymerase Chain Reaction on oropharyngeal rinse, non-invasive sampling and therefore probably less often positive and specific active infection. The investigators will develop a quantitative Polymerase Chain Reaction to identify a fungal load threshold number of copies / mL for diagnosing Pneumocystis jirovecii pneumonia with better positive predictive value.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Clinical or radiological indication for a broncho-alveolar lavage to search infectious agents including Pneumocystis jirovecii
* Patients with risk factors for developing a Pneumocystis jirovecii pneumonia : underlying malignancy (solid cancer, hematologic disease), organ transplant or hematopoietic stem cells, autoimmune disease or chronic inflammatory disease justifying immunosuppressive therapy (chemotherapy anticancer, immunomodulatory, biotherapy, corticosteroids) or patient treated with corticosteroids for more than a month or congenital immune deficiency or other causes of immunosuppression (excluding human immunodeficiency virus) at the discretion of the clinician,
* Informed consent given.

Exclusion Criteria:

* Patient human immunodeficiency virus positive
* Contraindication to the achievement of broncho-alveolar lavage,
* Contraindication to the achievement of a Oropharyngeal rinse (disorder of consciousness, swallowing disorder),
* Prophylaxis with cotrimoxazole or aerosol pentamidine,
* Empirical curative treatment with cotrimoxazole or other curative therapeutic alternative (pentamidine, atovaquone, dapsone, clindamycin-primaquine) started for more than 48 hours,
* Major person under legal protection (backup justice, trusteeship, guardianship), person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1250 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value of Polymerase Chain Reaction on oropharyngeal rinse | At the end of inclusion period (24 months)
  Definition of a numerical threshold from a multivariate analysis, for positioning the result of this test in combination with other clinical or laboratory parameters.

SECONDARY OUTCOMES:
Broncho-alveolar lavage Standardization | At the end of inclusion period (24 months)
  Definition of a quantitative threshold (number of copies / mL) for the interpretation of the Polymerase Chain Reaction on the broncho-alveolar lavage to estimate at best positive predictive value of Pneumocystis Polymerase Chain Reaction
Evaluation of serum dosage of β-1,3-D glucan | At the end of inclusion period (24 months)
  Definition of a positivity threshold to evoke a certain Pneumocystis jirovecii pneumonia, alone or in combination with Polymerase Chain Reaction.
Prevalence of genetic mutations of pneumocystis jirovecii | At the end of inclusion period (24 months)
  Analysis of the prevalence of mutations in the gene encoding the synthase dihydropteroate Pneumocystis jirovecii in patients with Pneumocystis jirovecii pneumonia or colonized and comparison with previous calculations Brittany and Picardy régions using a parametric test (t test) or nonparametric (Mann-test Whitney)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Robert-Gangneux, Md, PhD, Study Director — CHU Rennes
Locations (3):
- France (3):
  - CHU Amiens, Amiens
  - CHU Brest, Brest
  - CHU Rennes, Rennes